CLINICAL TRIAL: NCT06390709
Title: PREDICT Therapy Selection for JAK, T-cell, or IL-6 Inhibitor Therapies Using a Molecular Signature Response Classifier (PREDICT)
Acronym: PREDICT
Status: Recruiting | Type: Observational
Sponsor: Scipher Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: PREDICT-001
Record Dates: First submitted 2024-04-15; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JAK/T-cell/IL-6
  Interventions: Other: Lab Collection Only

INTERVENTIONS:
Other: Lab Collection Only — 2 Paxgene and 1 SST tubes will be collected at 2 timepoints throughout the study.

SUMMARY:
Prospective, multi-center-observational study conducted within the US, collecting patient samples for research and development to train, test, and validate precision medicine classifiers. These molecular signature response classifiers (MSRC) aim to predict response status to JAK, T-cell, and IL-6 inhibitor therapies in patients with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eighteen years of age, or older (≥18) at time of consent.
2. Patient must meet the criteria for RA as defined by the 2010ACR/EULAR classification at Visit 1 and documented by enrolling PI.
3. Patient has active RA, with moderate or high disease activity as confirmed by a CDAI score of >10 at Visit 1.
4. Patients must have a history of failure, contraindication, or intolerance to at least one csDMARD therapy.
5. Patient must be b/tsDMARD-naïve or TNFi-exposed prior to baseline visit only.
6. Patient must be initiating one of the following listed therapies (including biosimilars).

   1. JAK inhibitor therapy (only tofacitinib or upadacitinib)
   2. T-cell inhibitor therapy (abatacept)
   3. IL-6 inhibitor therapy (only tocilizumab)
7. Concomitant treatments are permitted per standard of care and are not limited to the following:

   a.csDMARD i.Methotrexate ii.Sulfasalazine iii.Leflunomide iv.Hydroxychloroquine b.Non-steroidal anti-inflammatory drugs c.Corticosteroids
8. Patient may participate in another observational study.
9. Patient is willing and able to complete the informed consent process and comply with all study procedures and visit schedule.

Exclusion Criteria:

1. Patient has previously participated in a Scipher Medicine study (NETWORK-004, AIMs in RA, DRIVE, or INFORM).
2. Patients who have been treated with an altMOA (non-TNFi therapy) therapy for RA prior to baseline (Visit 1).
3. Women who are known to be pregnant or breast-feeding or plan to get pregnant during the study duration.
4. Concurrent treatment with an investigational product or use of an investigational product within 28 days of Visit 1.
5. The use of RA therapies outside of an FDA approved indication.
6. Patient is currently receiving systemic antimicrobial treatment for viral, bacterial, fungal, or parasitic infection at the time of baseline visit (Visit 1).
7. Any known active, chronic, or recurrent invasive infection (e.g., listeriosis and histoplasmosis) and viral infection that, based on the Investigator's clinical assessment, makes the patient an unsuitable candidate for the study. This includes hepatitis B virus (HBV) or hepatitis C virus (HCV), recurrent or disseminated (even a single episode) herpes zoster, disseminated (even a single episode) herpes simplex, or human immunodeficiency virus (HIV).
8. Patient with any known active malignancy except non-melanoma skin cancer, localized prostate cancer treated with curative intent with no evidence of progression, low-risk or very low-risk (per standard guidelines) localized prostate cancer under surveillance/watchful waiting (without intent to treat),or carcinoma in situ of any type.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients with moderate or high disease activity and are eligible for treatment with a JAK, T-cell, or IL-6 inhibitor therapy who are either naïve to biologic and targeted synthetic DMARDs or TNFi-exposed.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of MSRC to predict the patients response | 6 months
  The rate of MSRC to predict the patients response status based on actual clinical disease activity measure at 6 months. Determine performance characteristics of the MSRC being developed, trained, and validated to predict a patient's response status to specific biologic or targeted therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- Medvin Clinical Research//Amicus Arthritis, Whittier, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT06390709/Prot_ICF_000.pdf